CLINICAL TRIAL: NCT01183702
Title: Analysis of Corneal Biomechanics Based Upon Central and Peripheral Corneal Thickness in Normal and Post Refractive Surgery Eyes
Brief Title: Corneal Biomechanics With Hydration in Normal and LASIK Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deb Grzybowski (Other)
Responsible Party: Sponsor-Investigator, Deb Grzybowski, Assistant Research Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2004H002
Record Dates: First submitted 2010-08-13; First posted 2010-08-18 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Laser Corneal Surgery
Keywords: LASIK vs. non-LASIK
MeSH Terms: interventions — Refractive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- non-LASIK (Active Comparator): These participants have NOT had LASIK surgery.
  Interventions: Other: No Intervention
- LASIK (Active Comparator): These participants have had LASIK surgery.
  Interventions: Procedure: LASIK surgery

INTERVENTIONS:
Procedure: LASIK surgery — Participants have received LASIK surgery and their eyes are healthy.
  Other Names: Refractive Surgery
  Arms: LASIK
Other: No Intervention — Participant has healthy eyes not altered by LASIK surgery.
  Other Names: Normal cornea; no refractive surgery
  Arms: non-LASIK

SUMMARY:
The research will utilize LASIK and non-LASIK populations to analyze the biomechanical differences between these corneas.

DETAILED DESCRIPTION:
The research will utilize LASIK and non-LASIK populations to analyze the biomechanical differences between these corneas. Subjects' corneas will be swelled with warmed, humidified nitrogen using modified diving goggles to assess structural changes due to a two hour swelling period. Subjects will be examined prior to swelling by a registered ophthalmologist to ensure that the cornea is healthy enough to undergo the swelling procedure. Pre-swelling and post-swelling data will be compared for parameters such as elasticity, density, thickness, axial and tangential curvature, hydration, and intraocular pressure in the central, paracentral, and peripheral regions. Analysis of pre-swelling and post-swelling data will allow for a better understanding of the structural changes created by LASIK. In addition, this project will allow for a better understanding of how common fluctuations in hydration levels affect normal corneal parameters as given by common devices in both populations to allow for corrections for more accurate measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy cornea without LASIK surgery as determined by a registered ophthalmologist.
* Healthy cornea with LASIK surgery as determined by a registered ophthalmologist.

Exclusion Criteria:

* Children under 18.
* Unhealthy cornea as determined by a registered ophthalmologist.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2004-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Corneal hydration (swelling) | Two hours

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M Grzybowski, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ophthalmology Department (Gowdy Field Building, 5th Floor), Columbus, Ohio, United States